CLINICAL TRIAL: NCT03004547
Title: Evaluation of Sodium Deposition in Soft Tissues of Patients with Kidney Disease and Its Association with Patient Symptomatology
Brief Title: Sodium Deposition in Soft Tissues of Patients with Kidney Disease
Status: Recruiting | Type: Observational
Sponsor: Chris McIntyre (Other)
Responsible Party: Sponsor-Investigator, Chris McIntyre, Professor of Medicine, UWO, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Organization: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Other Study IDs: 108765
Record Dates: First submitted 2016-12-16; First posted 2016-12-29 (Estimated); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Haemodialysis Complication
Keywords: Sodium; Soft Tissues

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — We will measure complete blood count, urea and electrolytes, magnesium, calcium, phosphate, liver function tests, clotting markers, cardiac biomarkers (Troponin T), 25-hydroxyVitamin D and 1,25-dihydroxyVitamin D, CRP, glucose, intact PTH, creatinine, cystatin C, and lactate.
  A portion of this blood sample will be sent to the laboratory on-site and the remaining portion will be for processed on-site and stored in the Kidney Clinical Research Unit, LHSC until the end of the study when endotoxin and uremic toxin measurement will be performed.
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (5):
- Chronic hemodialysis patients: Patients on standard in-centre 3 times a week hemodialysis
  Interventions: Other: Measuring sodium content
- Peritoneal dialysis patients: Patients on peritoneal dialysis
  Interventions: Other: Measuring sodium content
- Adult and paediatric patients with CKD stage 1-5: Patients with chronic kidney disease stage 1-5 (not dialysis dependent)
  Interventions: Other: Measuring sodium content
- Healthy adult and paediatric controls: Subjects without kidney disease
  Interventions: Other: Measuring sodium content
- Heart failure patients with and without renal dysfunction: Heart failure patients (atrial fibrillation etc ...) with and without renal dysfunction
  Interventions: Other: Measuring sodium content

INTERVENTIONS:
Other: Measuring sodium content — Sodium MRI measurement of sodium content in the tissues of all participants

SUMMARY:
Sodium (Na+) hemostasis is abnormal in CKD patients, and this element can be deposited in the skin, muscle, and skeleton - to cope with long term sodium loading. It is known that sodium stored in this non-osmotically active way, is profoundly inflammatory. Furthermore, inflammation has been associated with several uremic symptoms. The investigators will use novel Na+ MRI imaging to examine the Na+ deposition in the skin, muscle, and skeleton of five groups:1) chronic in-center hemodialysis patients, 2) chronic peritoneal dialysis patients, 3) adult and paediatric patients with CKD stage 1-5 and 4) heart failure patients with and without renal dysfunction 5) sex and age-matched healthy adult and paediatric controls. Additionally, they will investigate the association between sodium deposition in these tissues with uremic symptomatology and biochemical markers of metabolism.

DETAILED DESCRIPTION:
Kidneys have a key role in sodium hemostasis through their excretory function. In patients with chronic kidney disease (CKD), kidney function is impaired; thus, suggesting that sodium handling is abnormal in this setting with long-term sodium loading (from oral intake) and lack of adequate urinary excretion. Yet, sodium concentration needs to stay relatively constant to prevent fatal intra-cellular accumulation, which would result in cell injury and death. In hemodialysis patients, at least a part of this extra sodium is non-osmotically active and deposited in the skin, muscle, and skeleton.

Furthermore, it has become increasingly recognized that sodium (once accumulated in tissues) is directly pro-inflammatory, affecting the innate immune system by regulating the activity of macrophages in skin. This linkage between sodium and inflammation indicates a potential link between sodium deposition and uremic symptoms experienced by patients.

There have been no studies to date examining the sodium deposition in the skin, muscle, and skeleton of patients with different kidney function and renal replacement therapy.

This is a pilot study involving a single center recruiting patients from the prevalent maintenance hemodialysis, peritoneal dialysis , CKD stage 1-5, and heart failure populations of London, Ontario, compared to healthy controls. Once recruited, participants will undergo one study visit with the potential of up to two follow-up visits (on a non-dialysis day for hemodialysis patients). Participants will be followed for up to two years after the first study visit. Each session will include symptom questionnaires, the five times sit to stand and 60-second chair stand test (excluding all children), blood pressure and heart rate measurements, blood work (excluding healthy children and adolescents), urine sampling (excluding those on dialysis), an echocardiogram (excluding healthy controls), and an MRI scan of the lower leg detecting sodium content.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 6 years
* For patients on maintenance hemodialysis or peritoneal dialysis: more than 3 months duration of therapy
* For patients with CKD stage 1-5: CKD stage 1-5 and no indications to start dialysis
* For heart failure patients: with or without renal dysfunction
* For healthy controls: lack of kidney disease, heart failure, liver cirrhosis, and peripheral edema

For subsequent visits (must meet 1 of the below indicators):

* Change in dialysis prescription
* Change in renal replacement therapy modality
* Change in medication
* Parathyroidectomy
* Intervention added to or removed from dialysis (i.e. such as but not limited exercise, cooling, and ischemic preconditioning)

Exclusion Criteria:

* Pregnant, breastfeeding or intending pregnancy
* Unable to give consent or understand written information
* Contraindication to MRI study

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: We will recruit up to 400 participants; approximately 125 dialysis patients including 50 children/adolescents on dialysis, 200 patients with various stages of chronic kidney disease including heart failure patients and approximately 25 children/adolescents with chronic kidney disease, and 75 individuals with no kidney disease including approximately 25 healthy children/adolescents.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2018-03-05 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Na content in the skin, muscle and skeleton of five cohorts | 2 years

SECONDARY OUTCOMES:
Inflammatory Marker: CRP levels | 2 years
Uremic symptom scores among the different groups | 2 years
Liver function markers | 2 years
Liver damage markers (liver enzymes) | 2 years
cardiac markers (troponin) | 2 years
bone markers (ALP, vitamin D levels) | 2 years
Uremic toxin levels | 3-4 years
Endotoxin levels | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Christopher W McIntyre, PhD, MD, Principal Investigator — Western University, Canada
Locations (1):
- LHSC Regional Renal Care Program, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lemoine S, Salerno FR, Akbari A, McKelvie RS, McIntyre CW. Tissue Sodium Storage in Patients With Heart Failure: A New Therapeutic Target? Circ Cardiovasc Imaging. 2021 Nov;14(11):e012910. doi: 10.1161/CIRCIMAGING.121.012910. Epub 2021 Nov 16. PMID 34784242